CLINICAL TRIAL: NCT02921633
Title: Can Uptake of Childhood Influenza Immunisation in GP Practices be Increased Through Behavioural-insight Informed Changes to the Invitation Process?
Brief Title: Childhood Influenza Immunisation in General Practice Invitation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016_FluInvGP
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2016-09

CONDITIONS: Influenza, Human
Keywords: Immunization; Behavioural insights; Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention letter (Experimental): Centrally-sent behavioural-insight informed invitation letter.
  Interventions: Other: Intervention letter
- Control (No Intervention): No centrally-sent invitation letter.

INTERVENTIONS:
Other: Intervention letter
  Arms: Intervention letter

SUMMARY:
This study will investigate whether behaviourally informed changes to the invitation process can improve uptake of childhood influenza vaccine by two and three year olds at primary care.

DETAILED DESCRIPTION:
Previous research has shown that small changes to routine invitations/reminders to attend local health services informed by behavioural science can be used to increase a desired behaviour (e.g. uptake of health checks, reducing missed appointments).

This trial will determine whether an invitation letter, informed by behavioural insights and sent through a central system (Child Health Information System, CHIS), can increase uptake of childhood flu vaccine in primary care.

The trial will take place within the existing national childhood immunisation programme in the participating area in England. Randomisation will be clustered at the primary care practice level. Outcome data will be anonymised, routinely collected, individual-level influenza vaccine uptake data extracted from CHIS. For CHIS data validation purposes, practice-level vaccine uptake data reported through an alternative, routine system will be collected. Data will be collected on additional invitations/communications that primary care practices (in both the intervention and control arms) send to their patients. Cost data for the centralised letter will also be obtained.

The analysis will investigate the main effect of the intervention on uptake of the flu vaccination for all eligible children included in the trial. The model will include primary care practice and Clinical Commissioning Group effects to account for clustering. Secondary analysis will investigate the impact of such individual factors as age, immunisation history and socioeconomic status and practice-level factors (e.g. direct communication from practices) on uptake of the flu vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 2 years or 3 year olds at 31st August 2016
* Registered with a primary care practice in the participating area

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21786 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Influenza immunisation uptake | 4 months
  Immunisation uptake by eligible children (i.e. those aged 2 and 3 years on 31st August 2016) at primary care. Individual immunisation uptake data are routinely sent by primary care practices to the Child Health Information System. Anonymised uptake data will therefore be extracted for all eligible children from this system.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Chadborn, BSc MSc PhD, Principal Investigator — Public Health England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell-Jones R, Gold N, Bowen S, Bunten A, Tan K, Saei A, Jones S, MacDonald P, Watson R, Bennett KF, Chadborn T. Can uptake of childhood influenza immunisation through schools and GP practices be increased through behaviourally-informed invitation letters and reminders: two pragmatic randomized controlled trials. BMC Public Health. 2023 Jan 20;23(1):143. doi: 10.1186/s12889-022-14439-4. PMID 36670376